CLINICAL TRIAL: NCT03466645
Title: The Effectiveness of Vancomycin in Comarison With Cefazolin in Prevention of SSI After Craniotomy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Leila Dehghani, The effectiveness of vancomycin in comparison with cefazolin in prevention of SSI after craniotomy, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Isfahan University
Record Dates: First submitted 2018-03-09; First posted 2018-03-15 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2017-12

CONDITIONS: Elective Craniotomy-candidated Patients
Keywords: SSI; elective Craniotomy; Vancomycin; Cefazolin; Antibiotic
MeSH Terms: interventions — Vancomycin; Cefazolin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1st group, receiving vancomycin (Active Comparator): The 1st group receives vancomycin an hour before craniotomy
  Interventions: Drug: Vancomycin
- 2nd group, receiving cefazolin (Active Comparator): The 2nd group receives cefazolin an hour before craniotomy
  Interventions: Drug: Cefazolin

INTERVENTIONS:
Drug: Vancomycin — The 1st group receives vancomycin an hour before craniotomy
  Arms: 1st group, receiving vancomycin
Drug: Cefazolin — The 2nd group receives cefazolin an hour before craniotomy
  Arms: 2nd group, receiving cefazolin

SUMMARY:
Surgical-site infection is the most commonly reported nosocomial infection in patients undergoing surgery and 3rd most nosocomial infection in hospitalized patients. The SSI is associated with increases of length of hospitalization for 6 days and increases the hospital's cost by $ 300.

Because of these, prevention of SSI with appropriate antibiotic is essential.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years and above
* elective surgical patients
* No pre-surgery infection
* Do not use antibiotics before surgery
* Insensitivity to beta-lactam antibiotics

Exclusion Criteria:

* cranioplasty
* Failure to follow the patient
* The patient's unwillingness to continue participating in the research project
* Death of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
infection rate | Until 90 days after admission
  compare of infection rate in 2 groups

SECONDARY OUTCOMES:
length of hospitalization | Until 90 days after admission
  compare the length of hospitalization in 2 groups
raise of ESR & CRP | Until 90 days after admission
  compare the raise of ESR & CRP in 2 groups

CONTACTS AND LOCATIONS:
Locations (1):
- Isfahan university of medical science., Isfahan, Iran

IPD SHARING:
Plan to Share IPD: Undecided